CLINICAL TRIAL: NCT02888756
Title: A Phase IIa Randomized, Placebo Controlled, Double Blinded Study to Evaluate the Safety and Immunogenicity of iHIVARNA-01 in Chronically HIV-infected Patients Under Stable Combined Antiretroviral Therapy
Brief Title: iHIVARNA Clinical Trial in HIV Infected Individuals
Acronym: iHIVARNA-01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis did not show sufficient immunogenicity of IMP compared to placebo
Sponsor: Rob Gruters (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); IrsiCaixa (Other); Institute of Tropical Medicine, Belgium (Other); Vrije Universiteit Brussel (Other); Synapse bv (Industry); Asphalion (Unknown); eTheRNA immunotherapies (Industry); CR2O (Unknown); Hospital Clinic of Barcelona (Other); Germans Trias i Pujol Hospital (Other); Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor-Investigator, Rob Gruters, Workgroup leader, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: iHIVARNA phase II; 2016-002724-83 (EudraCT Number)
Record Dates: First submitted 2016-08-23; First posted 2016-09-05 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: Immunotherapy; mRNA; Lentivirus infection; Virus disease; Sexually transmitted disease; Immunodeficiency syndrome
MeSH Terms: conditions — HIV Infections; Lentivirus Infections; Virus Diseases; Sexually Transmitted Diseases; Immunologic Deficiency Syndromes | interventions — trimix

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iHIVARNA-01 (Experimental): Biological: 1200μg mRNA (900 μg HIV mRNA+300 μg TriMix mRNA) 3 vaccinations, two weeks interval
  Interventions: Biological: iHIVARNA-01; Biological: TriMix
- TriMix (Active Comparator): Biological: TriMix_300 μg TriMix mRNA 3 vaccinations, two weeks interval
  Interventions: Biological: TriMix
- Placebo (Placebo Comparator): Water for injection 3 vaccinations, two weeks interval
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: iHIVARNA-01 — Therapeutic vaccination, followed by treatment interruption
  Other Names: HIVACAT; TriMix
  Arms: iHIVARNA-01
Biological: TriMix — Therapeutic vaccination, followed by treatment interruption
  Arms: TriMix; iHIVARNA-01
Biological: Placebo — Therapeutic vaccination, followed by treatment interruption
  Arms: Placebo

SUMMARY:
iHIVARNA-01 is a novel therapeutic vaccine for the treatment of HIV-1-infected patients based on in vivo modification of DCs. It consists of HIVACAT-TriMix: mRNA encoding a mixture of APC activation molecules (CD40L, a constitutively active variant of TLR4 and CD70) and the HIV target antigens contained in HIVACAT to be administered through the intranodal route. iHIVARNA-01 aims to achieve the 'functional cure' of HIV infection, i.e. controlling viral replication in the absence of anti-retroviral therapy.

DETAILED DESCRIPTION:
Objective: To evaluate the safety and immunogenicity of iHIVARNA-01 as a new therapeutic vaccine in HIV infected patients.

Study design and duration: Phase IIa, multicentre double-blind placebo controlled intervention study. Each patient will be followed for 30 weeks. The study duration will be 38 weeks from inclusion of the first patient.

Sites: Erasmus MC, Rotterdam The Netherlands (sponsor), Hospital Clínic de Barcelona and Institut de Recerca de la Sida - Caixa, Barcelona, Spain, Instituut voor Tropische Geneeskunde Antwerp, Belgium and Vrije Universiteit Brussel/UZ Brussel, Belgium

Study population: Chronically HIV-1- infected patients under stable cART with plasma viral load (pVL) ≤ 50 copies/ml and stable CD4+ T-cell counts ≥ 450/μl, aged 18 years or above.

Sample size: after recruitment and screening, 70 patients will be included and randomized to one of the study-arms.

Intervention: One group (n=40) receives the HIVACAT-TriMix (300 microgram TriMix + 900 microgram HIVACAT) vaccine intranodally on three occasions with a two-week interval. One control group (n=15) receives TriMix only (300 microgram TriMix) and one group (n=15) receives saline intranodally on three occasions with a two-week interval. Two weeks after the last vaccination cART treatment will be interrupted. If plasma virus is detectable, cART will be re-initiated twelve weeks after treatment interruption. cART can always be re-initiated for medical reasons, as judged by the clinical investigator.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age;
2. Voluntarily signed informed consent;
3. Proven HIV-1 infection (with documented antibodies against HIV-1 and a detectable plasma HIV-1 RNA before initiation of therapy);
4. On stable treatment with cART regimen (antiretroviral therapy consisting of at least three registered antiretroviral agents) for at least 3 years;
5. Nadir CD4+ ≥ 350 cells/μl (up to 2 occasional determinations ≤ 350 cells/μl are allowed);
6. Current CD4+ cell count ≥ 450 cells/μl;
7. HIV-RNA below 50 copies/mL in the last 6 months prior to randomization, during at least two measurements (occasional so called 'blips' ≤ 500 copies/mL are permitted);
8. If sexually active, willing to use a reliable method of reducing the risk of transmission to their sexual partners during treatment interruption (including PrEP).

   1. For heterosexually active female, using an effective method of contraception with partner (combined oral contraceptive pill; injectable or implanted contraceptive; IUD/IUS; consistent record with condoms; physiological or anatomical sterility (in self or partner) from 14 days prior to the first vaccination until 4 months after the last vaccination.

For heterosexually active male, using an effective method of contraception with their partner from the first day of vaccination until 4 months after the last vaccination. -

Exclusion Criteria:

1. Treatment with non-cART regimen prior to cART regimen;
2. Previous failure to antiretroviral and/or mutations conferring genotypic resistance to antiretroviral therapy;
3. Non-subtype B HIV infection;
4. Active Hepatitis B virus and/or Hepatitis C virus co-infection;
5. History of a CDC class C event (see appendix A);
6. Pregnant female (screened with a positive pregnancy test), lactating or intending to become pregnant during the study;
7. Active malignancy ≤ 30 days (extended period on the clinical assessment of the investigator) prior to screening;
8. Active infection with fever (38°C or above) ≤ 10 days of screening and/or first vaccination;
9. Therapy with immunomodulatory agents (e.g. systemic corticosteroids), including cytokines (e.g. IL-2), immunoglobulins and/or cytostatic chemotherapy ≤ 90 days prior to screening. This does not include seasonal influenza, hepatitis B and/or other travel related vaccines;
10. Congenital, acquired or induced coagulation disorders, such as thrombocytopenia (thrombocytes < 150x109/L) and/or current use of anti-coagulant medication (e.g. coumarins, inhibitors of Xa); Usage of NSAIDs (including acetylsalicylic acid) is allowed, however it is advised to interrupt therapy 10 days ahead of vaccination;
11. Usage of any investigational drug ≤ 90 days prior to study entry;
12. An employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, or is a family member of an employee or the investigator Any other condition, which, in the opinion of the investigator, may interfere with the evaluation of the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob A Gruters, PhD, Principal Investigator — Erasmus Medical Center
Locations (5):
- Belgium (2):
  - Institute for Tropical Medicine, Antwerp
  - UZ Brussel, Brussels
- Erasmus MC, Rotterdam, Netherlands
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic, Barcelona

REFERENCES:
- [Derived] de Jong W, Aerts J, Allard S, Brander C, Buyze J, Florence E, van Gorp E, Vanham G, Leal L, Mothe B, Thielemans K, Plana M, Garcia F, Gruters R; iHIVARNA consortium. iHIVARNA phase IIa, a randomized, placebo-controlled, double-blinded trial to evaluate the safety and immunogenicity of iHIVARNA-01 in chronically HIV-infected patients under stable combined antiretroviral therapy. Trials. 2019 Jun 17;20(1):361. doi: 10.1186/s13063-019-3409-1. PMID 31208472
- See also: Description phase 1 clinical trial with iHIVARNA-01 — https://clinicaltrials.gov/ct2/show/NCT02413645

RESULTS

PARTICIPANT FLOW:
Period: Vaccination Period
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Started | 16 | 9 | 8
Completed | 16 | 9 | 8
Not Completed | 0 | 0 | 0
Period: Analytical Treatment Interruption
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Started (One participant did not start treatment interruption) | 15 | 9 | 8
Completed | 5 | 3 | 3
Not Completed | 10 | 6 | 5
Not completed — Physician Decision | 10 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iHIVARNA-01 | TriMix | Placebo | Total
Number analyzed (Participants) | 16 | 9 | 8 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 9 | 8 | 33
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 15 | 9 | 8 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 1 | 1 | 0 | 2
  Belgium | 6 | 3 | 3 | 12
  Spain | 9 | 5 | 5 | 19
CD4 T cell counts [Median (Inter-Quartile Range); unit: cells/microliter] | 793 [689 to 1041] | 708 [592 to 961] | 742 [679 to 918] | 769 [664 to 974]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: * Grade 3 or above local adverse event (pain, cutaneous reactions including induration).
  * Grade 3 or above systemic adverse event (temperature, chills, headache, nausea, vomiting, malaise, and myalgia).
  * Grade 3 or above other clinical or laboratory adverse event confirmed at examination or on repeat testing respectively.
  Any event attributable to vaccination leading to discontinuation of the immunisation regimen.
Time Frame: week 6
Measure: Count of Participants; unit: Participants
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Number analyzed (Participants) | 16 | 9 | 8
Participants | 0 | 0 | 0

2. Primary Outcome: Immunogenicity as Measured by Elispot
Description: Change from baseline immunogenicity as measured by ELISPOT at week 6 and 18, i.e. two weeks and 14 weeks after the last immunization compared to both control groups
Time Frame: week 6 and week 18
Measure: Mean (95% Confidence Interval); unit: delta log difference spot forming units
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Number analyzed (Participants) | 16 | 9 | 8
delta log difference spot forming units
  week 6 | -0.07 [-0.35 to 0.20] | 0.18 [-0.17 to 0.52] | 0.01 [-0.57 to 0.60]
  week 18 | -0.08 [-0.57 to 0.42] | -0.12 [-0.61 to 0.36] | 0.45 [-0.52 to 1.42]
Statistical Analysis 1: Comparison: iHIVARNA-01 vs TriMix vs Placebo; Analyzed for week 6, to provide statistical information for decision on execution of intracellular cytokine staining (ICS); Test type: Superiority; p = 0.14, Mixed Models Analysis

3. Secondary Outcome: Immunogenicity as Measured by Intracellular Cytokine Staining (ICS)
Description: HIV-specific CD4+ and CD8+ T cell responses after immunization by the number of poly-functional T cells as determined by intracellular cytokine staining, (ICS).
Time Frame: week 10, 18 and 30
Population: The data were not collected. In the protocol it was pre-specified, that ICS would not be done if Elispot results did not show immunogenicity of the study product. This analysis was not performed, because the results from the Elispot assay at the same time points showed no increase in the number of spot-forming units, also see primary outcome two.
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Time to Viral Rebound
Description: time until viral rebound (defined as two consecutive measurements of plasma viral load > 1000 copies/mL separated by at least 15 days) after discontinuation at week 6.
Time Frame: week 6-18
Population: One participant from the the iHIVARNA-01 group did not interrupt ART and therefor could not be analysed for time to viral rebound. Therefore the number in this group is 15 in stead of 16 at start of the trial.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Number analyzed (Participants) | 15 | 9 | 8
days | 50 [33 to 57] | 55.5 [43 to 77] | 58 [36 to 72]

5. Secondary Outcome: Change in Plasma Viral Load
Description: difference in log10 copies/ml plasma viral load in vivo after analytical treatment interruption (ATI, week 6-restart ART), compared to placebo WFI
Time Frame: week 6-18
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: log10 copies/ml
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Number analyzed (Participants) | 15 | 9 | 8
log10 copies/ml | -0.17 [-1.10 to 0.77] | -0.14 [-1.18 to 0.90] | 1.26 [0.21 to 2.31]

6. Secondary Outcome: Functional Cure
Description: proportion of patients with viral load below detectable level of 50 copies/mL in plasma after ATI, week 18
Time Frame: week 18
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Number analyzed (Participants) | 15 | 9 | 8
Participants | 0 | 0 | 0

7. Secondary Outcome: Primary Immune Response Against Vaccine
Description: Change in frequency of at least 0.7log10 HIV-specific T-cell responses between baseline and week 6
Time Frame: from baseline to week 6
Measure: Mean (95% Confidence Interval); unit: delta log spot forming units
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Number analyzed (Participants) | 13 | 7 | 6
delta log spot forming units | 0.01 [-0.56 to 0.57] | 0.17 [-0.47 to 0.81] | 2.65 [1.94 to 3.37]

8. Secondary Outcome: CD8 T Cell Mediated Viral Suppression
Description: The capacity of CD8 T cells to suppress virus production in HIV infected autologous CD4 T cells, after vaccination. For this purpose PBMC are isolated and separated in CD8 and CD4 T cells. CD4 cells are infected with HIV. Thereafter CD4 cells are co-cultured with pre-stimulated CD8 cells and the capacity to suppress virus production at different effector to target (E:T) ratios is measured, by the change of p24 Gag production. Pannus et al AIDS 2019, PMID: 30702513
Time Frame: week 4
Measure: Mean (95% Confidence Interval); unit: log(pg/ml)
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Number analyzed (Participants) | 10 | 9 | 5
log(pg/ml)
  stimulated (E:T) 2:1 | 0.15 [-0.69 to 0.99] | 0.22 [-0.73 to 1.16] | 0.18 [-0.48 to 0.85]
  Stimulated (E:T) 0.1:1 | -0.65 [-1.26 to -0.05] | -1.32 [-2.00 to -0.65] | 0.41 [-0.08 to 0.90]

9. Secondary Outcome: Proviral DNA Reservoir
Description: effect on reservoir as measured by changes in the proviral DNA copy numbers per million cells during and after immunization
Time Frame: day 0-90 (week 4, week 4 + 1 day and week 5 and week 6) and day 90-130 (week 18) and day >130 (week 30)
Measure: Mean (95% Confidence Interval); unit: delta log copies DNA /10E6 cel
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Number analyzed (Participants) | 16 | 9 | 8
delta log copies DNA /10E6 cel
  proviral DNA 0-90 days | -0.002 [-0.007 to 0.003] | -0.001 [-0.007 to 0.004] | 0.007 [0.003 to 0.011]
  proviral DNA 90-130 days | 0.004 [-0.010 to 0.019] | 0.004 [-0.013 to 0.020] | -0.003 [-0.015 to 0.008]
  proviral DNA >130 days | -0.001 [-0.007 to 0.005] | -0.002 [-0.010 to 0.006] | -0.003 [-0.007 to 0.002]

10. Secondary Outcome: Viral Immune Escape
Description: viral immune escape: change in % mutated epitopes from pre-cART to post-ATI
Time Frame: week 18
Population: data were not collected
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Transcriptomics
Description: host protein mRNA expression profiles in whole blood
Time Frame: week 6 and 18
Population: data were not collected
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Cell-associated RNA Viral Reservoir
Description: effect on reservoir as measured by changes in the intracellular viral RNA copy numbers per million cells during and after immunization
Time Frame: day 0-30 (week 4, week 4 + 1 day and week 5) and day 30-80 (week 6), 80-150 days (week 18) and >150 days (week 30)
Measure: Mean (95% Confidence Interval); unit: delta log copies RNA/ml
Arm/Group | iHIVARNA-01 | TriMix | Placebo
Number analyzed (Participants) | 16 | 9 | 8
delta log copies RNA/ml
  caRNA 0-30 days | -0.001 [-0.009 to 0.007] | -0.002 [-0.012 to 0.008] | -0.004 [-0.011 to 0.003]
  caRNA 30-80 days | -0.006 [-0.015 to 0.003] | -0.001 [-0.014 to 0.010] | 0.032 [0.024 to 0.040]
  caRNA 80-150 days | 0.002 [-0.008 to 0.012] | 0.003 [-0.008 to 0.015] | -0.016 [-0.024 to -0.008]
  caRNA >150 days | 0.002 [-0.008 to 0.011] | -0.001 [-0.012 to 0.010] | -0.004 [-0.011 to 0.003]

ADVERSE EVENTS:
Time Frame: 30 weeks
Arm/Group | iHIVARNA-01 | TriMix | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/16 | 0/9 | 1/8
Other Adverse Events (participants affected / at risk) | 16/16 | 9/9 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iHIVARNA-01 (N=16) | TriMix (N=9) | Placebo (N=8)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iHIVARNA-01 (N=16) | TriMix (N=9) | Placebo (N=8)
hypotensions (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (3) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 1 (1)
Chills (General disorders) | 2 (2) | 1 (2) | 1 (2)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 3 (5) | 2 (4)
influenza-like illness (General disorders) | 1 (2) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 1 (2)
Injection site pain (General disorders) | 3 (3) | 2 (3) | 2 (4)
Injection site puritis (General disorders) | 1 (1) | 0 (0) | 1 (2)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 3 (6) | 1 (1) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Tenderness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Urethritis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Burn-out syndrome (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Mental disoreder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatine-phospho kinase increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 6 (7) | 1 (1) | 4 (8)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Entercolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3)
Esophageal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythemia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Althragia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscles spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 2 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eyelid infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Furunkel (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastro enteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sexually transmitted disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Tonsillitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 4 (5) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limited number of subjects for statistical analysis due to early termination. There was an error in the study product, see https://insights.ovid.com/pubmed?pmid=31490219

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT02888756/Prot_SAP_000.pdf